CLINICAL TRIAL: NCT00254397
Title: Study of the Modulatory Activity of an LHRH-Agonist (Leuprolide) on Melanoma Peptide Vaccines as Adjuvant Therapy in Melanoma Patients
Brief Title: Melanoma Vaccine With Peptides and Leuprolide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004-0502
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Melanoma
Keywords: Melanoma; Uveal Melanoma; Peptide Vaccine; LHRH-agonist; Leuprolide; Lupron; MAGE-3 Peptide; MAGE-3; GP100 Peptide; Melanoma vaccines; Tumor fighting immune cells; T cells; Skin Cancer; Eye Cancer
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Skin Neoplasms; Eye Neoplasms | interventions — Leuprolide; Peptides; MAGEA3 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- gp100 + Leuprolide (Experimental): Group IA: HLA-A*0201 positive/HLA-DP4 negative treated with gp100 (1.0 ml subcutaneous injection in extremities) + Leuprolide (3-month 11.25 mg sustained-release formulation administrated intramuscularly then again 12 weeks later (2 injections)).
  Interventions: Drug: Leuprolide; Biological: GP100: 209-217(210M) Peptide
- gp100 - No Leuprolide (Experimental): Group IB: HLA-A*0201 positive/HLA-DP4 negative treated with gp100 (1.0 ml subcutaneous injection in extremities) - No Leuprolide
  Interventions: Biological: GP100: 209-217(210M) Peptide
- gp100 + MAGE-3 + Leuprolide (Experimental): Group IIA: HLA-A*0201positive/HLA-DP4 positive treated with gp100 (1.0 ml subcutaneous injection in extremities) + MAGE-3 (1.0 ml subcutaneous injection in extremities) + Leuprolide (3-month 11.25 mg sustained-release formulation administrated intramuscularly then again 12 weeks later (2 injections)).
  Interventions: Drug: Leuprolide; Biological: GP100: 209-217(210M) Peptide; Biological: MAGE-3 Peptide
- gp100 + MAGE-3 - No Leuprolide (Experimental): Group IIB: HLA-A*0201positive/HLA-DP4 positive treated with gp100 (1.0 ml subcutaneous injection in extremities) + MAGE-3 (1.0 ml subcutaneous injection in extremities) - No Leuprolide
  Interventions: Biological: GP100: 209-217(210M) Peptide; Biological: MAGE-3 Peptide

INTERVENTIONS:
Drug: Leuprolide — A 3-month 11.25 mg sustained-release formulation will be administrated intramuscularly at time 0, and approximately 12 weeks (2 injections).
  Other Names: Lupron Depot; Lupron
  Arms: gp100 + Leuprolide; gp100 + MAGE-3 + Leuprolide
Biological: GP100: 209-217(210M) Peptide — 1.0 ml subcutaneous injection in extremities.
Biological: MAGE-3 Peptide — 1.0 ml subcutaneous injection in extremities.
  Other Names: MAGE-3
  Arms: gp100 + MAGE-3 + Leuprolide; gp100 + MAGE-3 - No Leuprolide

SUMMARY:
The goal of this clinical research study is to learn if the drug leuprolide will increase the level of immune cells in your body. Researchers will also want to know if this drug given together with melanoma vaccines (gp100 and MAGE-3) can improve the ability of tumor fighting immune cells (T cells) to fight melanoma cells.

Primary Objective:

1. To compare the tumor-specific immune responses to melanoma-specific peptide vaccines, gp100 and MAGE-3 in the presence or absence of a luteinizing hormone-releasing hormone (LHRH) agonist-Leuprolide, in patients with stage IIb and III melanoma, uveal melanoma or stage IV melanoma that the metastatic lesion(s) has been surgically removed.

Secondary Objectives:

1. To evaluate the kinetics of enhanced thymic activity measured by TREC analysis and flow cytometric analysis following sex hormone ablation by Leuprolide in melanoma patients.
2. To assess whether there are significant differences in overall quality of life (QOL) between patients receiving Leuprolide to those not receiving leuprolide.

DETAILED DESCRIPTION:
This study uses vaccines named gp100 or MAGE-3 to immunize patients with melanoma. The type of melanoma they will be used for contains a protein that is also found in the vaccines. These vaccines are designed to stimulate immune cells, also called T cells, to recognize and kill melanoma cells. Leuprolide will be studied to determine whether it will (is designed to) improve your response to the vaccine.

If you are eligible for this treatment, you will be assigned to one of the two groups that either receive one vaccine or two different vaccines, depending on your tissue type (either gp100 vaccine alone or gp100 and MAGE-3 vaccines). A small amount of the vaccine(s) will be injected under your skin to test your body's immune response to the vaccines. The size of the skin reaction will be measured at 48-72 hours. This skin test will be done before you receive any vaccine, at 6 months, and at 12 months, if possible.The participant and/or participant's family will be given detailed verbal and written instructions on how to measure any reaction to the skin tests. A data sheet and ruler (cm/mm) will be given to the participant.

You will then be randomly assigned (as in the toss of a coin) to one of 2 treatment groups. Participants in one group will receive leuprolide with the vaccine(s). Participants in the other group will not receive leuprolide. Which group you are assigned to will depend partially on your age.

If you are assigned to receive leuprolide injection, you will also have a bone mineral density test to check on the strength of your bones.

Before the treatment starts, you will be asked to answer a questionnaire about your quality of life and sexual functioning. Then at 3 months and 12 months of treatment, you will be asked again to answer the same questionnaire. It should take about 20 minutes each time to finish the questionnaire.

The vaccines will be injected in the skin every 3 weeks for a total of 48 weeks. Those patients in Group I will receive 32 injections of peptide, whereas those patients in Group II will receive 64 injections of peptide over a 48 week period. If you are assigned to receive leuprolide, then leuprolide will be injected in the muscle at the beginning of the study and at 12 weeks, for a total of 2 additional injections. Both the vaccine and leuprolide injections will be given each time at the melanoma outpatient clinic at M. D. Anderson.

Blood (about 4 teaspoons) will be taken at 6 weeks, 12 weeks, then every 12 weeks up to 48 weeks, or at any time if your tumor starts to grow back. Researchers will use this blood to find out how well your immune cells are working to fight your tumor cells.

At around 24 weeks and 48 weeks into treatment, your will have CT scans of the chest, abdomen and pelvis to check on the status of your disease. At around 24 weeks, if you are receiving leuprolide and had an abnormal bone mineral density test before the treatment, you will also have the second bone mineral density test to check on the strength of your bones.

You may be taken off study if your disease gets worse or intolerable side effects occur. If you are taken off study, you will be asked to have repeat scans and a physical exam, including blood (about 4 tablespoons) for routine tests.

Following the first 48 week treatment period, you will be evaluated every 3 months for one year, every 4 months for one year, every 6 months for one year, and then once a year from then on if clinically feasible.

You will have an MRI/CT of the brain, chest, abdomen and pelvis to check on the status of your disease. If your disease gets worse or intolerable side effects occur, you will be taken off study.

Blood (about 4 tablespoons) will be drawn for routine lab tests. An additional 4 tablespoons of blood will be drawn at each follow-up visit to determine how long the t-cell counts remain high.

This is an investigational study. Gp100 and MAGE-3 vaccines are experimental and authorized for research use only. Leuprolide is approved in treating prostate cancer patients and other gynecological diseases, but is not approved for treatment of melanoma. Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. HLA-A *0201 positive
2. Patients >/= 18 years old with histologically documented diagnosis of stage IIb-IV melanomas and are clinically rendered free of disease after surgery
3. Uveal melanoma patients following definitive treatment of radiation therapy and/or enucleation.
4. Karnofsky Performance Scale >/= 60%.
5. White Blood Count (WBC) >/= 3000/mm^3.
6. Platelet count >/= 90,000mm^3.
7. Serum creatinine </= 2.0mg/dl.
8. Serum alanine aminotransferase (ALT) </= 3 times upper limit of normal(ULN))
9. Total bilirubin equal or less than 2 times upper limit of normal (ULN)), except for patient with Gilbert's syndrome who must have a total bilirubin less than 3.0mg/dl.
10. Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
11. Negative pregnancy test by serum or urine b-HCG test for women who have menstruation in the past 12 months and without sterilization surgery.
12. Unless surgically sterile by bilateral tubal-ligation or vasectomy of partner(s), the subject agrees to continue to use a barrier method of contraception throughout the study such as: condom, or diaphragm, or sponge plus spermicide. Abstinence is an acceptable form of birth control.

Exclusion Criteria:

1. Prior systemic therapy (including immunomodulate agents), radiation or surgery requiring general anesthesia for melanoma within 28 days of starting study treatment.
2. Autoimmune diseases.
3. Concurrent systemic or inhaled steroid therapy.
4. Any form of active primary or secondary immunodeficiency.
5. History of immunization with gp100 or MAGE-3.
6. Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, surgically treated Stage I or II cancer from which the patient is currently in complete remission (at least for 5 years), or any other cancer from which the patient has been disease-free for 5 years.
7. Received a Luteinizing hormone-releasing hormone (LHRH) agonist within the past 5 years.
8. Use of oral contraceptive, hormone replacement therapy or androgen preparations.
9. Hypersensitivity to gonadotropin-releasing hormone analogues.
10. Active systemic infections requiring intravenous antibiotics.
11. Lactating women or women planning lactation during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hwu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of Recruitment Period: November 8, 2005 to August 11, 2009. All participants recruited the University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | gp100 + Leuprolide | gp100 - No Leuprolide | gp100 + MAGE-3 + Leuprolide | gp100 + MAGE-3 - No Leuprolide
Started | 10 | 6 | 37 | 45
Completed | 4 | 5 | 18 | 20
Not Completed | 6 | 1 | 19 | 25
Not completed — Disease Progression | 4 | 1 | 16 | 23
Not completed — Non-Compliant | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | gp100 + Leuprolide | gp100 - No Leuprolide | gp100 + MAGE-3 + Leuprolide | gp100 + MAGE-3 - No Leuprolide | Total
Number analyzed (Participants) | 10 | 6 | 37 | 45 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 27 | 31 | 72
  >=65 years | 1 | 1 | 10 | 14 | 26
Age, Continuous [Median (Full Range); unit: years] | 48.5 [29 to 72] | 43.5 [26 to 71] | 55 [20 to 85] | 54 [21 to 84] | 53 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 11 | 18 | 35
  Male | 5 | 5 | 26 | 27 | 63
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 37 | 45 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With T-cell Response to Peptide Vaccine
Description: Reactivity to the gp100 peptide in each participant defined as >10 tetramer positive cells per 10^4 CD8+ T-cells as determined by the tetramer analysis at 3 months following initial vaccine. Number of participants with response as defined reported.
  The primary end point of this clinical study was the comparison of tumor-specific immune responses to melanoma-specific peptide vaccines, gp100 and MAGE-3 in the presence or absence of Leuprolide.
  Gp209-2M/HLA-A*0201 tetramers that are commercially available employed to analyze levels of gp209-2M specific CD8+ cytolytic T cells. The levels of peptide/ HLA-A*0201 tetramer between participants' peripheral blood mononuclear cells (PBMCs) with Leuprolide injection and without Leuprolide injection compared.
Time Frame: At 3 months following initial vaccine.
Population: Although all participants did not receive all doses of the vaccine due to tumor progression and other reasons, if samples were available after two or more vaccinations, analyses were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | gp100 + Leuprolide | gp100 - No Leuprolide | gp100 + MAGE-3 + Leuprolide | gp100 + MAGE-3 - No Leuprolide
Number analyzed (Participants) | 7 | 4 | 26 | 33
Participants | 6 | 1 | 12 | 19

2. Secondary Outcome: Most Frequent and Most Serious Participant Adverse Events During Vaccine Treatment for Overall Study
Description: Summary of most frequent adverse events collected study wide during vaccine treatment period using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Time Frame: Baseline up to 48 weeks during vaccine treatment
Population: Although our immunologic analysis was based on participants HLA type in order to determine reactivity against particular peptides, all participants received vaccines with or without leuprolide. Therefore, in assessing toxicity we analyzed participants within these two groups.
Measure: Number; unit: occurences
Groups:
- gp100 + No Leuprolide: HLA-A*0201 positive/HLA-DP4 negative treated with gp100 (1.0 ml subcutaneous injection in extremities)
Arm/Group | gp100 + Leuprolide | gp100 + No Leuprolide
Number analyzed (Participants) | 47 | 51
occurences
  Elevated Creatinine | 1 | 0
  Hyperglycemia | 1 | 0
  Cardiac troponin T | 1 | 0
  Cardiac Ischema | 1 | 0
  Fatigue | 15 | 7
  Hypotension | 1 | 0
  Ruptured lumbar disc | 1 | 0
  Possible Metastatic Lung Nodule | 1 | 0
  Cellulitis | 1 | 0
  Cerebral Ischemia | 1 | 0
  Cardiac Ischemia/stent | 1 | 0
  Atrial fibrillation | 2 | 0
  Multiple Allergic Reactions | 1 | 0

3. Secondary Outcome: Number of Participants Experiencing Adverse Events by Maximum Grade Within Different Arms
Description: Maximum Grade reported for participant adverse events. collected study wide during vaccine treatment period using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Time Frame: Baseline up to 48 weeks during vaccine treatment
Population: Only 91 participants' data was available for classification in analysis.
Measure: Number; unit: participants
Arm/Group | gp100 + Leuprolide | gp100 - No Leuprolide | gp100 + MAGE-3 + Leuprolide | gp100 + MAGE-3 - No Leuprolide
Number analyzed (Participants) | 10 | 4 | 36 | 41
participants
  Grade 4-Life threatening or disabling | 0 | 0 | 1 | 0
  Grade 3-Severe | 2 | 0 | 0 | 3
  Grade 2-Moderate | 5 | 2 | 21 | 10
  Grade 1-Mild | 2 | 2 | 7 | 24

4. Secondary Outcome: Summary of Adverse Events by Grade/Relationship
Description: Summary of adverse events( AE) collected during vaccine treatment period using Common Terminology Criteria for Adverse Events v3.0 (CTCAE). Grade 0-Sign/symptom within normal limits, Grade 1-Mild AE, Grade 2-Moderate AE, Grade 3-Severe AE, Grade 4- Life threatening or disabling AE.
Time Frame: Baseline up to 48 weeks during vaccine treatment
Measure: Number; unit: occurences
Arm/Group | gp100 + Leuprolide | gp100 - No Leuprolide | gp100 + MAGE-3 + Leuprolide | gp100 + MAGE-3 - No Leuprolide
Number analyzed (Participants) | 10 | 6 | 37 | 45
occurences
  Grade 4, Unspecified Relationship | 0 | 0 | 1 | 0
  Grade 3, Possible | 1 | 0 | 0 | 1
  Grade 3, Probable | 1 | 0 | 0 | 0
  Grade 3, Unrelated | 0 | 0 | 0 | 1
  Grade 3, Unspecified Relationship | 0 | 0 | 0 | 1
  Grade 2, Definite | 5 | 0 | 11 | 0
  Grade 2, Possible | 3 | 1 | 19 | 3
  Grade 2, Probable | 5 | 0 | 3 | 1
  Grade 2, Unlikely | 0 | 0 | 2 | 3
  Grade 2, Unrelated | 3 | 1 | 1 | 4
  Grade 2, Unspecified Relationship | 8 | 1 | 16 | 7
  Grade 1, Definite | 21 | 4 | 61 | 50
  Grade 1, Possible | 22 | 6 | 103 | 74
  Grade 1, Probable | 13 | 3 | 53 | 56
  Grade 1, Unlikely | 16 | 4 | 25 | 38
  Grade 1, Unrelated | 15 | 3 | 45 | 36
  Grade 1, Unspecified Relationship | 29 | 7 | 61 | 37
  Grade 0, Possible | 1 | 0 | 0 | 0
  Grade 0, Probable | 2 | 0 | 0 | 0
  Grade 0, Unlikely | 0 | 0 | 2 | 0
  Grade 0, Unrelated | 0 | 0 | 0 | 0
  Grade 0, Unspecified Relationship | 2 | 0 | 5 | 13

ADVERSE EVENTS:
Time Frame: Participants evaluated every 6 weeks up to 48 weeks during the vaccine treatment phase of the study. Active study participation period: November 2005 to October 2010 (last participant off study).
Description: Although our immunologic analysis was based on patient HLA type in order to determine reactivity against particular peptides, all patients received vaccines with or without leuprolide. Therefore, in assessing toxicity we analyzed patients within these two groups.
Groups:
- gp100, Leuprolide, MAGE-3: HLA-A*0201 positive/HLA-DP4 negative treated with gp100 (1.0 ml subcutaneous injection in extremities) with/without Leuprolide (3-month 11.25 mg sustained-release formulation administrated intramuscularly then again 12 weeks later (2 injections)); with/without MAGE-3 (1.0 ml subcutaneous injection in extremities)
- gp100 + No Leuprolide: HLA-A*0201 positive/HLA-DP4 negative treated with gp100 (1.0 ml subcutaneous injection in extremities) without Leuprolide; with/without MAGE-3 (1.0 ml subcutaneous injection in extremities)
Arm/Group | gp100, Leuprolide, MAGE-3 | gp100 + No Leuprolide
Serious Adverse Events (participants affected / at risk) | 3/47 | 3/51
Other Adverse Events (participants affected / at risk) | 47/47 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | gp100, Leuprolide, MAGE-3 (N=47) | gp100 + No Leuprolide (N=51)
Cardiac Ischemia/ Infarction (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Neutrophils Elevated (Blood and lymphatic system disorders) | 0 | 1 — Absolute neutrophil count (ANC)
Pain (Head/Headache) (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | gp100, Leuprolide, MAGE-3 (N=47) | gp100 + No Leuprolide (N=51)
Allergic rhinitis (Immune system disorders) | 5 | 0
Bone development abnormal (Musculoskeletal and connective tissue disorders) | 9 | 0
Dizziness (Nervous system disorders) | 19 | 2
Fatigue (General disorders) | 15 | 7
Fever of unknown origin (Infections and infestations) | 9 | 3
Gynecomastia (Reproductive system and breast disorders) | 15 | 0
Headache (Nervous system disorders) | 25 | 1
Hot Flashes (Endocrine disorders) | 31 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 1
Impotence (Reproductive system and breast disorders) | 15 | 0
Infections (Infections and infestations) | 6 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 16 | 16
Insomnia (General disorders) | 22 | 2
Libido (Reproductive system and breast disorders) | 19 | 0
Lymphopenia (Infections and infestations) | 5 | 0
Mood Alteration (Nervous system disorders) | 46 | 0
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 9 | 2
Myalgia (General disorders) | 13 | 7
Neuropathy:Sensory (Nervous system disorders) | 45 | 2
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 30 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 12 | 10
Rash (Skin and subcutaneous tissue disorders) | 26 | 0
Vaginitis (Reproductive system and breast disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No